CLINICAL TRIAL: NCT04526912
Title: A Proof of Concept Study of the Safety and Efficacy of VIB7734 for the Treatment and Prevention of Acute Lung Injury (ALI) in Patients With SARS-CoV-2 Infection
Brief Title: Treatment and Prevention of Acute Lung Injury (ALI) in Patients With COVID-19 Infection
Acronym: ALI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study met predefined futility criteria for efficacy endpoints.
Sponsor: Viela Bio (Industry)
Responsible Party: Sponsor
Organization: Viela Bio (acquired by Horizon Therapeutics) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIB7734.P1.S2
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Acute Lung Injury
Keywords: pneumonia; COVID-19; SARS-Cov-2; acute respiratory disease
MeSH Terms: conditions — Acute Lung Injury; Pneumonia; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIB7734 Dose (Experimental): Participants will receive a single subcutaneous dose of VIB7734.
  Interventions: Drug: VIB7734
- Placebo (Placebo Comparator): Participants will receive a single subcutaneous dose of placebo (saline) matched to single dose of VIB7734.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIB7734 — Single subcutaneous dose
  Arms: VIB7734 Dose
Drug: Placebo — Intravenous single dose matched to VIB7734.
  Arms: Placebo

SUMMARY:
The study aims to assess the potential benefit and evaluate the safety and tolerability of a single subcutaneous (SC) dose of VIB7734 in hospitalized patients with documented infection of severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) with pulmonary involvement. Subjects will be administered a single dose of VIB7734 injected under the skin, assessed for efficacy for 28 days and followed for an additional 42 days.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study intended to assess the potential benefit and evaluate the safety and tolerability of a single subcutaneous (SC) dose of VIB7734 in hospitalized patients with documented infection of severe acute respiratory syndrome coronavirus 2 (SARS CoV-2) with pulmonary involvement. Efficacy will be assessed during the 28 days following a single administration of VIB7734. Safety will be assessed for 10 weeks following dosing. The pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of VIB7734 in patients with confirmed SARS-CoV-2 infections will also be assessed.

ELIGIBILITY:
Key Inclusion Criteria:

* Hospitalized with coronavirus disease 2019 (COVID-19) pneumonia confirmed by World Health Organization criteria.
* Oxygen saturation ≤ 94% at room air or arterial partial pressure of oxygen/fraction of inspired oxygen < 300 mm Hg and > 200 mm Hg.
* Negative influenza test.
* Lymphocyte counts < 10^3/μL and the presence of at least one of the following markers of hyperinflammation within 1 day prior to VIB7734 administration:

  * Elevated high sensitivity C-reactive protein (hsCRP) > 50 mg/L
  * Ferritin > 500 ng/mL
  * Lactate dehydrogenase (LDH) > 300 U/L
  * D-dimers > 500 ng/mL

NOTE: Other protocol defined inclusion criteria apply

Key Exclusion Criteria:

* Respiratory failure requiring mechanical ventilation.
* In the opinion of the Investigator, progression to mechanical ventilation or death is imminent and inevitable within the next 24 hours.
* Valid Do Not Intubate (DNI) or Do Not Resuscitate (DNR) order.
* Anticipated duration of hospital stay < 72 hours.
* History of allergy or hypersensitivity reaction to any component of the IP.
* Participation in another clinical study with an IP within 4 weeks prior to Day 1 or within 5 half-lives of the IP, whichever is longer. (Participation in COVID-19 antiviral or antimalarial trials may be permitted after discussion with the Medical Monitor).
* Liver cirrhosis or liver failure.
* Known human immunodeficiency virus infection.
* Known hepatitis B or known hepatitis C infection in the absence of a history of curative therapy.
* Known or suspect active or latent tuberculosis infection.
* Active bacterial, fungal, viral, or other infection (besides COVID-19).
* Clinically significant cardiac disease within 6 months.
* History of severely impaired respiratory function at baseline (not related to COVID-19) based on requirement for home oxygen of > 4 L/min or based on other medical history known to the Investigator.
* History of cancer within 12 months of enrollment.
* Receipt of chemotherapy, biologic immunomodulators (including JAK inhibitors), or immunosuppressive therapies within 8 weeks of enrollment, or receipt of rituximab or other B cell-depleting mAb therapy within 6 months.

NOTE: Other protocol defined exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieve treatment success through Day 28, defined as avoidance of death and critical illness | Day 1 (Baseline) through Day 28
  Critical illness is defined by respiratory failure (requiring any of the following: endotracheal intubation, oxygen delivered by high flow nasal cannula, non-invasive positive pressure ventilation, extracorporeal membrane oxygenation or clinical diagnosis of respiratory failure) or shock (systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg, or requiring vasopressors)

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent fatal and life-threatening SAEs, Treatment-emergent Serious Adverse Events | Day 1 (Baseline) through Day 70
  Defined as measure of safety
Change in safety laboratory parameters | Day 1 (Baseline) through Day 70
  Safety evaluation via review of labs (white blood cell (WBC) with differential counts, hemoglobin, platelet count, liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], and total bilirubin levels), serum chemistry, cardiac troponin coagulation markers (prothrombin time [PT], partial thromboplastin time [PTT], D dimer, fibrinogen), and urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Illei, MD, PhD, MHS, Study Director — Vice President, Clinical Development Lead
Locations (1):
- Research Site, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No